CLINICAL TRIAL: NCT02597985
Title: Prehabilitation to Improve Functional and Clinical Outcomes in Patients Undergoing Transcatheter Aortic Valve Replacement: TAVR-FRAILTY Trial
Brief Title: Prehabilitation to Improve Functional and Clinical Outcomes in Patients With Aortic Stenosis
Acronym: TAVR-FRAILTY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mandeep Singh, Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-004180
Record Dates: First submitted 2015-10-26; First posted 2015-11-05 (Estimated); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Aortic Stenosis
Keywords: Frailty
MeSH Terms: conditions — Aortic Valve Stenosis; Frailty | interventions — Preoperative Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prehabilitation (Active Comparator): Will receive 4 weeks of supervised exercised prescription before they undergo TAVR and will monitor and record, improvement if any, in the short-term physical performance battery score
  Interventions: Other: Prehabilitation
- Usual care (Placebo Comparator): Will receive usual care
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Prehabilitation — Supervised exercise training intervention will include three sessions per week for four weeks at a Mayo Clinic system cardiac rehabilitation facility. The Rochester, Minnesota Cardiac Rehabilitation Program will provide guidance and oversight. Modes of aerobic exercise will include treadmill walking (the primary mode of training) supplemented with non-weight-bearing activities such as stationary cycling and combination arm/leg recumbent exercise (NuStep device), as needed. Intensity will be set using Borg Perceived Exertion Scale (RPE) ratings of 12-14 (somewhat hard), keeping patients below the threshold for more than mild angina.
  Arms: Prehabilitation
Other: Usual Care
  Arms: Usual care

SUMMARY:
Transcatheter aortic valve replacement (TAVR) is a treatment alternative among high-risk elderly with aortic stenosis, however, mortality remains high. Fifty percent of patients undergoing TAVR exhibit frailty, a syndrome associated with poor survival. It is unknown whether interventions to improve frailty before TAVR (prehabilitation) will improve outcomes after TAVR. This study plans to evaluate whether simple cardiac exercise interventions to improve physical performance before TAVR improves outcomes after TAVR.

ELIGIBILITY:
Inclusion criteria:

* Eligibility for TAVR
* SPPB<9
* Able to exercise
* Able to come for follow-up visits
* Able to give informed consent

Exclusion criteria:

* New York Heart Association (NYHA) Class III/IV congestive heart failure (CHF)
* Presyncope or syncope as presentation
* Acute coronary syndrome
* Unable to exercise
* Dementia
* Sustained ventricular arrhythmia
* Stroke with neurological deficit
* Advanced Parkinson's
* Participated in an exercise program

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-10; Primary Completion 2019-06-17 (Actual); Study Completion 2019-09-10 (Actual)

PRIMARY OUTCOMES:
Change in Score on short physical performance battery (SPPB) test | Baseline, approximately 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mandeep Singh, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials